CLINICAL TRIAL: NCT00233961
Title: Peripheral Blood Stem Cell Mobilization With Filgrastim in Patients With Chronic Myeloid Leukemia in Cytogenetic Response
Brief Title: G-CSF in Stimulating Peripheral Stem Cells for Autologous Stem Cell Transplant in Treating Patients With Chronic Phase Chronic Myeloid Leukemia in Complete Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441128; CPMC-AAAA9963
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — Filgrastim

INTERVENTIONS:
Biological: filgrastim

SUMMARY:
RATIONALE: Giving colony-stimulating factors, such as G-CSF, helps stem cells move from the bone marrow to the blood so they can be collected and stored until transplant.

PURPOSE: This phase I trial is studying the side effects of G-CSF in stimulating peripheral stem cells for autologous stem cell transplant in treating patients with chronic phase chronic myeloid leukemia in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and safety of harvesting adequate numbers of CD34-positive peripheral blood stem cells using filgrastim (G-CSF) in patients with chronic phase chronic myeloid leukemia in complete cytogenetic remission.
* Determine the safety of temporarily discontinuing treatment with imatinib mesylate and using G-CSF during the harvesting procedure, in terms of the percentage of Philadelphia chromosome (Ph)-positive cells before and after stem cell harvest, in these patients.

OUTLINE: Patients receive filgrastim (G-CSF) and then undergo apheresis for up to 5 days.

After completion of apheresis, patients resume treatment with imatinib mesylate off study. Patients may later undergo autologous peripheral blood stem cell transplantation, when deemed necessary.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic phase chronic myeloid leukemia

  * In complete cytogenetic remission, confirmed by bone marrow biopsy within the past month
* Has been receiving imatinib mesylate for ≥ 3 months* NOTE: *Imatinib mesylate is held during the study harvesting procedure
* No myelofibrosis on bone marrow ≥ 3+
* Ineligible for or refused allogeneic stem cell transplantation

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,000/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Adequate hepatic function for stem cell transplantation

Renal

* Adequate renal function for stem cell transplantation

Cardiovascular

* Adequate cardiovascular function for stem cell transplantation

Pulmonary

* Adequate pulmonary function for stem cell transplantation

Other

* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent biologic therapy

Chemotherapy

* More than 4 weeks since prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy

Surgery

* No concurrent surgery

Other

* No other concurrent experimental therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of harvesting chronic myeloid leukemia (CML) patients in continuous complete remission (CCR) by adequate CD34+ stem cell numbers post-harvest

SECONDARY OUTCOMES:
Effect of discontinuation of imatinib during harvesting by cytogenetic evaluation post-harvest

CONTACTS AND LOCATIONS:
Overall Officials: Gwen L. Nichols, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York, United States